CLINICAL TRIAL: NCT04239131
Title: A Prospective Study About the Sensitization Patterns to Insects as Food Source in Patients With House Dust Mite Allergy Based on Clinical History, Skin Prick Tests and in Vitro Tests
Brief Title: Prospective Study About Sensitization Pattern to Insects as Food Source in Patients With House Dust Mite Allergy
Acronym: InFood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: InFood2020
Record Dates: First submitted 2020-01-06; First posted 2020-01-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hypersensitivity, Food
MeSH Terms: conditions — Food Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Patients (Other): It is a single arm study. Skin prick testing and laboratory Tests are carried out on all patients in the same way
  Interventions: Other: Skin prick test

INTERVENTIONS:
Other: Skin prick test — a Skin prick test is planned in all patients

SUMMARY:
Patients allergic to seafood and/or sensitized to Tropomyosin of Skin Prick tests SPT or crustacean origin will may be also be sensitized to edible insects. Aim of the study is to evaluate whether patients allergic to seafood and/or sensitized to Tropomyosin of SPT or crustacean origin may be more often be sensitized to edible insects used as food source.

DETAILED DESCRIPTION:
House dust mite allergy is a common problem in Europe. In addition to inhalant allergies sensitization to mites can be related to food allergy namely seafood. Insects are also widespread food sources in many regions of the world.

In this study skin testing and laboratory tests are planned in patients with known house dust mite allergy to evaluate a possible sensitization to insects. Patients must also complete a questionnaire. A drug therapy or other intervention is not planned.

Aim of the study is to evaluate whether patients allergic to seafood and/or sensitized to Tropomyosin of SPT or crustacean origin may be more often be sensitized to edible insects used as food source.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 < x < 70
* House dust mite sensitization with or without sensitization to seafood
* Subject is capable of giving informed consent
* Signed informed consent

Exclusion Criteria:

* Use of antihistamines, systemic corticosteroids during testing and within three days (antihistamines) or two weeks (corticosteroids) prior to testing
* Use of immunosuppressive agents
* History of cancer except for treated basal cell or spinal cell carcinoma of the skin
* Active or recurrent bacterial, fungal or viral infection at the time of enrollment, including patients with evidence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection, active or untreated latent tuberculosis.
* Female patients of childbearing potential who are pregnant or breast feeding or planning a pregnancy during the duration of the trial and/or not practicing acceptable birth control for the duration of the trial
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrollment into the current study,
* Enrollment of the investigator, his/her family members, employees and other dependent persons,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Presence/absence of insect sensitization among seafood/Tropomyosin-sensitized patients versus patients with house dust mite sensitization alone | 1 week
  Sensitization (+/-)

SECONDARY OUTCOMES:
Sensitization pattern in insect sensitized patients in comparison between seafood-sensitized versus non-seafood-sensitized patients | 1 week
  Sensitization (+/-)
Sensitization pattern in seafood sensitizes patients in comparison between insect-sensitized versus non-insect-sensitized patients | 1 week
  Sensitization (+/-)
Sensitization pattern in insect sensitized patients in comparison between resident and immigrant populations in Switzerland | 1 week
  Sensitization (+/-)
Sensitization pattern in seafood sensitized patients in comparison between resident and immigrant populations in Switzerland | 1 week
  Sensitization (+/-)
Frequency of sensitization to the various insect allergens | 1 week
  Sensitization (+/-)
Description of possible cross reactions between seafood and insect allergens | 1 week
  Sensitization (+/-)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, MD, Principal Investigator — Universitätsspital Zürich
Locations (1):
- Allergy Unit,University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No